CLINICAL TRIAL: NCT03551145
Title: Patient Perception and Clinical Efficacy of Geistlich Mucograft® vs. Autologous Connective Tissue Graft for the Treatment of Peri-implantitis: Multi-centre Randomized Clinical Trial
Brief Title: Patient Perception and Clinical Efficacy of a Collagen Matrix for the Treatment of Peri-implantitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: PerioCentrum Research (Other)
Responsible Party: Principal Investigator, Prof. Elena Figuero, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16/502-P
Record Dates: First submitted 2018-05-09; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Multi-centre randomized clinical trial (2 centres) with the duration of 102 weeks for the evaluation of efficiency on the new collagen xenograft (Muco-Graft®) in comparison to the autologous connective tissue graft for the augmentation of keratinized mucosa and gaining hygienic access to the implants diagnosed with peri-implantitis
Who Masked: Investigator, Outcomes Assessor
Masking Description: The examiners will be blinded. Envelopes will be prepared by a research assistant not involved as clinician or examiner. The clinicians involved will have no access to the data collection sheets or the group allocation, whilst the examiners will have no access to the patients' treatment notes or group allocation. The examiners will be blinded with regards to the participant treatment assignments. The measures will include no access to the dental records as to which treatment has been assigned. The patients are not to reveal their treatment assignment to the examiners. Unblinding is expected when patients present with adverse outcomes during the course of the study, e.g., emphysema.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acellular collagen matrix (Experimental): In a test group, partial thickness-flap will be elevation will be performed, in order to create the vascular recipient bed for the randomized graft. Implant surface will be treated with ultrasound device, glycine powder and implantoplasty in case of the exposure of the rough surface. Acellular collagen matrix will be adapted and suture to the vascular bed.
  Interventions: Other: Acellular collagen matrix
- Autogenous free gingival graft (Active Comparator): In a control group, partial thickness-flap will be elevation will be performed, in order to create the vascular recipient bed for the randomized graft. Implant surface will be treated with ultrasound device, glycine powder and implantoplasty in case of the exposure of the rough surface. Free gingival graft will be harvested from the zone of the posterior palate, and then adapted and sutured to the vascular bed.
  Interventions: Other: Autogenous free gingival graft

INTERVENTIONS:
Other: Acellular collagen matrix — 3D collagen matrix consists of the collagen porcine type I and III
  Arms: Acellular collagen matrix
Other: Autogenous free gingival graft — Autogenous graft harvested from the posterior palate
  Arms: Autogenous free gingival graft

SUMMARY:
This is a multi-centre, randomized clinical trial which evaluates the efficiency of the collagen xenograft (Muco-Graft®) in comparison to the autologous connective tissue graft for the augmentation of keratinized mucosa and gaining hygienic access to the implants diagnosed with peri-implantitis.

DETAILED DESCRIPTION:
Nowadays, there is not enough evidence that evaluates the patient's perception of utilizing the soft tissue substitutes in comparison to the autologous connective tissue graft for the augmentation of the keratinized mucosa and gain of hygienic access to the implants with infectious pathology and with minimum or absent keratinized mucosa.

Therefore, the aim of the study is to evaluate the change of clinical parameters of peri-implant health and the patient perception of the procedure for augmentation of the keratinized tissues around dental implants with peri-implantitis.

The hypothesis is that collagen matrix of porcine origin is associated with lower patient morbidity, in comparison with autologous connective-tissue graft, when used for the augmentation of the keratinized tissues around endosseous dental implants with infectious pathology and with minimum or absent KT mucosa.

A sample 48 patients will be recruited basing upon the diagnosis of peri-implantitis and absent or insufficient peri- implant mucosa. 1 month after the non-surgical treatment, surgical procedure will be performed.

Peri-implant clinical and radiographic parameters, as well as patient perception of the therapy provided, will be evaluated before and at various stages (up to 52 weeks) after the surgical intervention. Also, change of vestibulum depth will be analyzed, as well as the time spent for the procedure measured.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent after the detailed information on the study.
* Adults aged at least 18 years old.
* Candidates for receiving augmentation of the peri-implant keratinized mucosa.
* Presence of the implant diagnosed with peri-implantitis (radiographic bone loss > 2 mm, with a probing depth > 5 mm, bleeding and/or suppuration (Lang et al., 2011)).
* Absent or insufficient keratinized peri-implant mucosa (<2 mm).

Exclusion Criteria:

* General contraindications for the dental/surgical treatment;
* Inflammatory or autoimmune disease of the oral cavity;
* Implant with radiographic intraosseous defects more than 3 mm;
* Smokers > 10 cig/day;
* Allergy to collagen or analgesics/anti-inflammatory non-steroid drugs;
* History of cancer in various parts of the body which required radiotherapy or chemotherapy during the last 5 years;
* Radiotherapy of the head or neck in the last 5 years;
* Actual medication with immunosuppressors, bisphosphonates or high doses of corticosteroids;
* Pregnant or lactating women;
* Women in fertile age, who do not use effective methods of contraception;
* Participants of other studies of biomedical investigation during the last 24 weeks before initiation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in width of keratinized peri-implant mucosa | Baseline, 0, 1, 2, 4, 12, 26 and 52 weeks
  Measured by periodontal probe (UNC-15), as mm of keratinized mucosa in the midbuccal portion of the implant of interest

SECONDARY OUTCOMES:
Bleeding on probing | Baseline, 0, 1, 2, 4, 12, 26 and 52 weeks
  Measured as presence or absence (binary value) of bleeding 10 seconds after probing with the periodontal probe in 6 point around each implant
Probing depth | Baseline, 0, 1, 2, 4, 12, 26 and 52 weeks
  Measured by periodontal probe (UNC-15) in millimeters in 6 points around each implant, and defined as a distance from the mucosal margin to the bottom of the peri-implant pocket
Recession | Baseline, 0, 1, 2, 4, 12, 26 and 52 weeks
  Measured by periodontal probe (UNC-15) in millimeters in 6 points around each implant, and defined as a distance from the implant platform to the mucosal margin
General satisfaction by the treatment | 0, 1, 2, 4, 12, 26 and 52 weeks
  Measured by a questionnaire, using the visual analogue scale, in values from 0 to 100
Duration of surgery | after completion of surgical intervention
  Measured by the electronic timer in minutes, starting from the moment of first incision and ending with a last suture
Vestibulum depth | Baseline, 0, 1, 2, 4, 12, 26 and 52 weeks
  Measured in mm by a periodontal probe, as a distance from the mucosal margin to the point of greatest concavity of the mucobuccal fold

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Univesity Complutense, Madrid, Madrid, Spain